CLINICAL TRIAL: NCT01776255
Title: Healthy Children, Strong Families: American Indian Communities Preventing Obesity
Acronym: HCSF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2012-0578; 1R01HL114912-01 (NIH)
Record Dates: First submitted 2013-01-16; First posted 2013-01-28 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Overweight; Lifestyle; American Indian
MeSH Terms: conditions — Obesity; Overweight | interventions — Child Restraint Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Children, Strong Families (first) (Experimental): Healthy Children, Strong Families intervention (first). This is a series of monthly educational tool kits mailed to primary caregivers for use with the participating child. This arm crosses over to receive the Child Safety in Year 2.
  Interventions: Behavioral: Healthy Children, Strong Families; Behavioral: Child Safety
- Child Safety (first) (Active Comparator): A series of 12 monthly newsletters and providing education on child safety mailed to primary caregivers. This Arm crosses over to receive the Healthy Children, Strong Families intervention in Year 2.
  Interventions: Behavioral: Healthy Children, Strong Families; Behavioral: Child Safety

INTERVENTIONS:
Behavioral: Healthy Children, Strong Families — Healthy Children, Strong Families is a series of 13 "lessons" mailed to primary caregivers of preschool aged children that provide education and activities related to obesity prevention. The lessons cover topics related to nutrition, physical activity, stress, sleep, and the home environment. Lessons include printed materials and small items (for example, an apple sectioner) that support activities in the lessons. Social support components via a monitored Facebook group and approximately semiweekly text messages sent to caregivers are included. The intervention spans 1 year.
Behavioral: Child Safety — The Child Safety intervention is an active control condition consisting of monthly two-page newsletters covering various topics relevant to child safety such as choking, car safety seats, bike and pedestrian safety. The intervention spans 1 year.

SUMMARY:
Healthy Children, Strong Families-2 (HCSF-2) is a family focused early childhood intervention which addresses the growing problem of childhood obesity in American Indian communities. The study works with six rural and urban American Indian communities across the US to test the ability of the intervention to increase adoption of healthy lifestyles and to reduce the prevalence of obesity among preschool aged American Indian children and their primary caregivers - creating healthier children, healthier families and healthier communities. Our primary hypothesis is that children and their primary caregivers who receive the HCSF-2 intervention will have better obesity related outcomes than those who do not receive HCSF-2.

DETAILED DESCRIPTION:
Intervention

The Healthy Children, Strong Families-2 (HCSF-2) intervention consists of monthly mailed healthy lifestyle lessons (13 lessons) which will be dose enhanced with social networking support (cell-phone coaching with instant text messages and Facebook connections), as well as new intervention elements-stress and sleep. Social networking was chosen due to its widespread and ease of use, adaptability and potential for sustainability in the community.

HCSF-2 is based on our hypothesis that working with children and their primary caregivers/parent to assist them in making healthy lifestyle changes is necessary to prevent excessive weight gain and risk of later lifestyle related chronic disease. Investigators will work with families at a critical time in their young child's physical and emotional development to encourage appropriate healthy lifestyle behaviors.

This study will expand on our previous research to test the HCSF-2 intervention in a larger, more geographically and socially diverse sample of AI communities. The study also enhances the prior methodology through the inclusion of a social networking component. This research will address four key gaps in obesity prevention studies: families with preschool age children, social networking support, stress and sleep. Moreover, to our knowledge, this study will be the first family-based obesity intervention project for both rural and urban AI families. The potential impact of this study is high; if successful, this study will not only provide quantitative evidence of the effectiveness of the intervention but it will also give other investigators validated tools and procedures to collaboratively engage AI communities in health behavior change.

Year 1, families will be randomized to start in the HCSF-2 intervention or an active control (mailed child safety newsletters). Then, in Year 2, intervention change will occur, such that HCSF-2 intervention families will receive the control safety lessons plus continued HCSF-2 social networking, while control families will now receive the full HCSF-2 intervention.

For example, families will be randomly assigned to begin in one of the two arms - denoted here as the HCSF-2 intervention (Phase A) or Child Safety intervention (Phase B).

During the HCSF-2 intervention (Phase A) families will receive a monthly mailing with information about nutrition and physical activity, screen time, sleep and stress management. Families will also be invited to participate in a private Facebook group and will begin receiving wellness coaching text messages from the study.

During the Child Safety intervention (Phase B) families will receive a monthly mailing with information about safety topics such as car safety, water safety, poisoning and home safety.

After one year, families will flip into the second phase until the two year study period is complete. Families who began in Phase A will continue to receive wellness coaching text messages and have access to the private Facebook group. Families who began in Phase B will not receive wellness coaching text messages or have access to the private Facebook group until the flip into Phase A at the start of year two.

This staggered enrollment design, chosen in conjunction with the participating communities, maximizes the contribution of each participating family, avoids the negative attitudes that would occur with a wait-list only control and ensures all families receive the intervention as desired by the participating tribal sites.

This is a multi-site trial with up to six possible participating communities. Two sites will become active at the beginning of the intervention with remaining sites becoming active (and being added to the IRB protocol) at roughly 1 year intervals.

A local site coordinator will be hired at each participating site. The local site coordinator will be responsible for recruiting participants, and conducting data collection visits. Site coordinators may also send wellness coaching text messages and post content to the private Facebook group.

The UW program coordinator will be responsible for screening participants for eligibility, administering 24-hour dietary recalls by phone, mailing HCSF-2 curriculum materials and Child Safety materials, managing the entry and storage of study data, sending results letters to participants and supporting the community site coordinators.

Methods

Investigators will partner with 6 diverse rural and urban AI communities nationally to conduct a 2-arm staggered-enrollment randomized trial of an enhanced version of the HCSF intervention (HCSF-2) vs. active control (Child Safety intervention) in a 2-year design with outcomes measured at 0, 6, 12, 18 and 24 months. At the end of year 1, control families will receive HCSF-2, and HCSF-2 families will receive the control intervention with continued HCSF-2 social network support. Communities will work with us to enhance the family-focused HCSF-2 intervention to include novel methods of delivery (mailed lessons with social networking/cell phone text coaching) and two less-studied obesity determinants-sleep and stress-to increase impact and sustainability.

Outcomes

Primary outcomes will be body fat as assessed by child Body Mass Index z-score (zBMI) and adult Body Mass Index (BMI). Secondary outcomes include adult and child waist circumference, fruit/vegetable (FV) and added sugar intake, TV/screen time, activity, sleep, home environment changes, adult psychosocial factors (stress/depression) and social network use.

Investigators will also identify key mediators of the effect of HCSF-2 on obesity and health behaviors. We hypothesize that modifiable behavior changes in children and caregivers, adult self-efficacy, social support and home environment changes are important mediators of the effect of the intervention on obesity and other outcomes. Investigators will develop and test exploratory mixed-effects regression models to investigate mediation on the path from HCSF-2 to weight reduction.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregiver with a 2-5 year old child
* 2-5 year old child with a caregiver
* Caregiver has a working cell phone and is willing to receive regular text messages as part of study participation
* Caregiver lives within feasible travel distance of data collection site and willing to come for data collection visits at 0, 6 months, 12 months, 18 months and 24 months
* Willingness to be randomized to one of two groups with the understanding that all participants will receive all components of the intervention, randomization simply determines the order in which materials are received
* Valid mailing address where participant can receive mail and packages
* Basic English fluency and literacy sufficient for understanding the intervention materials and completing questionnaires

Exclusion Criteria:

* Adults with no children or whose only children are younger than 2 or older than 5
* Children younger than 2 or older than 5 years of age
* No cell phone or unwilling to receive regular text messages as part of study participation
* Lives beyond feasible travel distance of data collection sites AND/OR planning on moving out of the area within a two year period
* Child has major physical or behavioral disorder (e.g. failure to thrive, severe autism) that would seriously impact study participation
* No valid mailing address
* Unwillingness to accept random allocation to study arm
* Spouse/partner of another caregiver-child pair who is living in same home & who has already enrolled (e.g. only one adult-child pair per household may be enrolled)

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Change in child adiposity from baseline measured via BMI z-score | Enrollment, 6 months, 12 months, 18 months, 24 months
  BMI z-score is obtained by computing the BMI weight (in kg)/height (in m)*height (in m). BMI is then converted to a z-score based on US national norms for gender and age in months provided
Change in adult adiposity from baseline measured via BMI | Enrollment, 12 months, 24 months
  Adult BMI is computed from weight (in kg) divided by height (in m) squared

SECONDARY OUTCOMES:
Change in child adiposity from baseline measured via waist circumference | Enrollment, 6 months, 12 months, 18 months, 24 months
  Waist circumference (in cm) is measured with a plastic measuring tape
Change in adult adiposity from baseline measured via waist circumference | Enrollment, 12 months, 24 months
  Waist circumference (in cm) is measured with a plastic measuring tape
Change in child fruit and vegetable consumption from baseline | Enrollment, 12 months, 24 months
  Child fruit and vegetable consumption measured via a 13-item questionnaire completed by the primary caregiver that is based on questions contained in the 2010 National Youth Physical Activity and Nutrition Survey published by the Centers for Disease Control and Prevention
Change in adult fruit and vegetable consumption from basline | Enrollment, 12 months, 24 months
  Adult fruit and vegetable consumption is measured with a 30-item questionnaire published by the National Cancer Institute.
Change in amount of child screen time from basline | Enrollment, 12 month, 24 month
  Amount of time spent watching TV, videos, video games, and computer are assessed via 8 items on a questionnaire completed by primary caregiver.
Change in amount of adult screen time from basline | Enrollment, 12 month, 24 month
  Amount of time spent watching TV, videos, video games, and computer are assessed via 8 items on a questionnaire.
Change in amount of child physical activity from baseline | Enrollment, 12 months, 24 months
  Child physical activity is measured via primary caregiver's responses to the 8 items on the Netherlands Physical Activity Questionnaire.
Change in amount of adult physical activity from basline | Enrollment, 12 months, 24 months
  Adult physical activity is measured via the 4 item Godin physical activity questionnaire.
Change in child sleep pattern from basline | Enrollment, 12 months, 24 months
  Primary caregivers complete a 6-question sleep questionnaire on sleep timing (weekday and weekend bedtime and awakening)and sleep duration in hours as well as sleep latency for both themselves and the participating child.
Change in home environment from basline | Enrollment, 12 months, 24 months
  Primary caregivers complete a 24 item questionnaire pertaining to the availability of supports and family routines relevant to physical activity and nutrition.
Change in adult Readiness to Change from basline | Enrollment, 6 months, 12 months, 18 months, 24 months
  Primary caregivers complete a 7 item questionnaire pertaining to readiness to change behaviors relevant to obesity.
Change in adult SF-12 scores from basline | Enrollment, 12 months, 24 months
  Primary caregivers complete a 12-item questionnaire that poses questions about their perception of their physical and emotional well being.
Stress questionnaire | Enrollment, 12 months, 24 months
  Primary caregivers complete a 10-item questionnaire pertaining to perceptions of global areas of stress.
Change in adult sleep pattern from basline | Enrollment, 12 months, 24 months
  Primary caregivers complete a 6-question sleep questionnaire on sleep timing (weekday and weekend bedtime and awakening)and sleep duration in hours as well as sleep latency for both themselves and the participating child.

OTHER OUTCOMES:
Parent 24 hour dietary recalls | Enrollment, 12 month, 24 month
  24 hour dietary recalls (Nutrition Data Services) will be conducted on primary caregiver and child to provide validation of results obtained in the fruit and vegetable questionnaires. Child recalls will be conducted via caregiver proxies.
Cultural Identity Scale | Enrollment, 12 months, 24 months
  Adult caregivers complete a 6-item measure of acculturation specific to American Indians that yields a general score for involvement in traditional culture. This measure is not expected to change as a result of the study but is being collected as a potential moderating variable.
Child Safety Survey | 12 months, 18 months
  An 8-item questionnaire is completed by primary caregivers receiving the Child Safety active control intervention to assess their attention the the newsletters and obtain their feedback.
HCSF Participant Survey | 12 months, 18 months
  A 26-item survey assess participant involvement and gathers feedback on the HCSF intervention and materials.
All Participant Exit Survey | 24 months
  A 30-item survey requests feedback on many aspects of the project.
Child 24 hour dietary recalls | Enrollment, 12 month, 24 month
  24 hour dietary recalls (Nutrition Data Services) will be conducted on primary caregiver and child to provide validation of results obtained in the fruit and vegetable questionnaires. Child recalls will be conducted via caregiver proxies.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra K Adams, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - White Earth Child Care Program, White Earth, Minnesota
  - Blackfeet Nation, Browning, Montana
  - First Nations HealthSource, Albuquerque, New Mexico
  - Seneca Nation, Irving, New York
  - Menominee Tribe of Wisconsin, Keshena, Wisconsin

REFERENCES:
- [Background] Adams AK, LaRowe TL, Cronin KA, Prince RJ, Wubben DP, Parker T, Jobe JB. The Healthy Children, Strong Families intervention: design and community participation. J Prim Prev. 2012 Aug;33(4):175-85. doi: 10.1007/s10935-012-0275-y. PMID 22956296
- [Background] Jobe JB, Adams AK, Henderson JA, Karanja N, Lee ET, Walters KL. Community-responsive interventions to reduce cardiovascular risk in American Indians. J Prim Prev. 2012 Aug;33(4):153-9. doi: 10.1007/s10935-012-0277-9. PMID 22983753
- [Background] LaRowe TL, Wubben DP, Cronin KA, Vannatter SM, Adams AK. Development of a culturally appropriate, home-based nutrition and physical activity curriculum for Wisconsin American Indian families. Prev Chronic Dis. 2007 Oct;4(4):A109. Epub 2007 Sep 15. PMID 17875253
- [Derived] Tomayko EJ, Webber EJ, Cronin KA, Prince RJ, Adams AK. Use of Text Messaging and Facebook Groups to Support the Healthy Children, Strong Families 2 Healthy Lifestyle Intervention for American Indian Families. Curr Dev Nutr. 2021 May 17;5(Suppl 4):32-39. doi: 10.1093/cdn/nzaa110. eCollection 2021 Jun. PMID 34222765
- [Derived] Rink E, Knight K, Ellis C, McCormick A, FireMoon P, Held S, Webber E, Adams A. Using Community-Based Participatory Research to Design, Conduct, and Evaluate Randomized Controlled Trials with American Indian Communities. Prev Chronic Dis. 2020 Nov 12;17:E143. doi: 10.5888/pcd17.200099. PMID 33180688
- [Derived] Tomayko EJ, Prince RJ, Cronin KA, Kim K, Parker T, Adams AK. The Healthy Children, Strong Families 2 (HCSF2) Randomized Controlled Trial Improved Healthy Behaviors in American Indian Families with Young Children. Curr Dev Nutr. 2018 Nov 16;3(Suppl 2):53-62. doi: 10.1093/cdn/nzy087. eCollection 2019 Aug. PMID 31453428
- [Derived] Grant VM, Tomayko EJ, Prince RJ, Cronin K, Adams A. Understanding Correlates of Physical Activity in American Indian Families: The Healthy Children Strong Families-2 Study. J Phys Act Health. 2018 Nov 1;15(11):866-873. doi: 10.1123/jpah.2017-0584. Epub 2018 Oct 19. PMID 30336717
- [Derived] Tomayko EJ, Mosso KL, Cronin KA, Carmichael L, Kim K, Parker T, Yaroch AL, Adams AK. Household food insecurity and dietary patterns in rural and urban American Indian families with young children. BMC Public Health. 2017 Jun 30;17(1):611. doi: 10.1186/s12889-017-4498-y. PMID 28666476